CLINICAL TRIAL: NCT06252961
Title: Randomized, Double-blind Trial Evaluating the Safety and Efficacy of a 3- or 5- Day Course of Levamisole 2.5 mg/kg in Subjects With Loa Loa Microfilaremia
Brief Title: A 3- to 5-day Clinical Trial of Levamisole in Loiasis Infected Subjects
Acronym: STOP-FiLAR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Programme National de Lutte contre l'Onchocercose, Republic of the Congo (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocole128
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Loiasis
Keywords: Onchocerciasis; Filariasis; Levamisole
MeSH Terms: conditions — Loiasis; Onchocerciasis; Filariasis | interventions — Levamisole

STUDY DESIGN:
Intervention Model Description: A 3-group, randomized, double-blind, parallel clinical trial:
  * Levamisole 2.5 mg for 3 days (followed by 2 days placebo),
  * Levamisole 2.5 mg for 5 days,
  * Placebo for 5 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Levamisole 3 days (Experimental): Participants randomized in this arm will receive 3 days of levamisole 2.5mg/kg, followed by 2 days of placebo
  Interventions: Drug: Levamisole 3 days
- Levamisole 5 days (Experimental): Participants randomized in this arm will receive a 5-day course of levamisole 2.5mg/kg
  Interventions: Drug: Levamisole 5 days
- Placebo (Placebo Comparator): Participants randomized in this arm will receive 5 days of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levamisole 3 days — Levamisole for 3 days (2,5 mg/kg) then placebo for 2 days
  Arms: Levamisole 3 days
Drug: Levamisole 5 days — Levamisole for 5 days (2,5 mg/kg)
  Arms: Levamisole 5 days
Drug: Placebo — Placebo for 5 days
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of a 3- and 5-day course of levamisole (2.5 mg/kg) in management of loiasis microfilaremia.

DETAILED DESCRIPTION:
Onchocerciasis and loiasis are parasitic diseases caused by Onchocerca volvulus and Loa loa, respectively.

Onchocerciasis is endemic in 31 African countries, parts of South America, and Yemen, affecting around 37 million people, while loiasis is present in Central Africa, infecting approximately 15 million individuals. Both diseases are associated with severe complications and increased mortality.

African countries have implemented mass drug administration (MDA) programs using ivermectin to combat onchocerciasis. However, co-endemic loiasis poses challenges due to the risk of severe adverse events. Current strategies involve alternative treatments and chemoprophylaxis to accelerate onchocerciasis elimination. The project aims to evaluate the use of levamisole as an alternative treatment.

This project will assess the safety and efficacy of administering levamisole for 3 and 5 days to reduce Loa microfilarial density. Previous research demonstrated the safety of a single dose of levamisole but indicated the need for longer treatment regimens to achieve a significant reduction in Loa microfilarial density. The project aims to test whether 3- and 5-day levamisole regimens induce an acceptable safety profile and a stronger reduction in Loa microfilarial density.

ELIGIBILITY:
Inclusion Criteria:

* Consent informed, written, signed and dated
* Women or men aged 18 to 65 years inclusive
* Carrier of L. loa microfilaremia
* Body weight ≥ 40 kg in women and ≥ 45 kg in men; and less than 90 kg
* In good health, as determined by medical questionnaire and general clinical examination
* Absence of acute or chronic infection :

Exclusion criteria

* Participation in any study other than a purely observational study, within the 4 weeks preceding this study (determined by the theoretical date of the first administration of levamisole or placebo)
* Any vaccination within 4 weeks previous to this study
* Infection requiring treatment in the 10 days previous to this study, as determined by the anamnesis during the medical interview (e.g. pulmonary infection , digestive or skin infection; with or without antibiotic treatment)
* Treatment with clozapine, phenothiazines, sulfasalazine, carbamazepine, synthetic antithyroid drugs, ticlopidine, cimetidine, and gold salts: whether it was long-term treatment, or treatment given as a single dose 10 days before the start of treatment for the clinical trial (precaution with regard to the risk of agranulocytosis of immuno-allergic or toxic origin)
* Known immunosuppressive pathology (by self-report)
* Past or present history of neurological (including epilepsy) or neuropsychiatric disease
* History of agranulocytosis
* Use of cocaine or other drugs of abuse in the 72 hours preceding administration of the trial treatment, as determined by history during the medical interview
* Any condition, in the opinion of the investigator, that exposes the subject to undue risk
* Known intolerance to levamisole
* Subjects who donated blood in the previous 8 weeks to study entry, with a standard volume (> 500 mL)
* On clinical examination: symptoms, physical signs or laboratory findings suggestive of systemic disorders, including disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other abnormalities that could interfere with the interpretation of trial results. The physician may then give a favorable or unfavorable opinion on the participant's inclusion.
* Ivermectin and/or levamisole taken in the last six months; and/or mebendazole or albendazole taken in the last month
* Pregnant and/or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2024-09-18 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Tolerance of multiple doses of levamisole 2.5 mg/kg in individuals with Loa loa microfilaremia | During the treatment (5 days) and 2 weeks after
  The proportions of adverse reactions and severe adverse reactions between the three arms of study will be compared, as well as between each interventional arm versus placebo, using appropriate comparative tests A multivariate analysis may be envisaged to assess the influence of age, gender and the presence or absence of M. perstans on the proportion of AEs

SECONDARY OUTCOMES:
Efficacy of multiple doses of levamisole 2.5 mg/kg on Loa loa microfilaremia | From Day 3 after the first dose to Day 30 after the first dose
  Microfilaremia reduction rates will be compared between arms at Day 3, Day 5, Day 7, Day 15 and Day 30. The proportions of subjects who had reduced their microfiflaremia by at least 80% at D3, D5, D7, D15 and D30 will be compared Finally, a multivariate analysis could be carried out to assess the influence of age, gender and the presence or absence of M. perstans on the reduction of the microfilaremia.

CONTACTS AND LOCATIONS:
Overall Officials: Jéremy CAMPILLO, PharmD PhD, Study Director — Institut de Recherche pour le Développement (IRD); François MISSAMOU, MD, Principal Investigator — Programme National de Lutte contre l'Onchocercose (PNLO)
Locations (2):
- Republic of the Congo (2):
  - Supervisor, Sibiti, Komono
  - General Supervisor, Sibiti, Mokassi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chesnais CB, Hemilembolo MC, Sahm BA, Toutin F, Djeutassong E, Nga-Elomo N, Cuer B, Ntsiba-N'Goulou MA, Pakat M, Pion SDS, Missamou F, Boussinesq M, Campillo JT. Safety and efficacy of 3- and 5-day regimens of levamisole in loiasis: a randomized, placebo-controlled, double-blind clinical trial. Nat Commun. 2025 Jul 4;16(1):6191. doi: 10.1038/s41467-025-61479-6. PMID 40615414